CLINICAL TRIAL: NCT05971862
Title: An Open-label, Multi-center, Dose-escalation and Dose-finding, Phase I Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of SKI- G-801 as Monotherapy in Patients With Advanced Solid Tumors
Brief Title: A Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of SKI-G-801 in Patients With Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Oscotec Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: OSCO-P1302
Record Dates: First submitted 2023-06-29; First posted 2023-08-02 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- SKI-G-801(Denfivontinib) 100mg QD (Experimental): Administered orally
  Interventions: Drug: SKI-G-801
- SKI-G-801(Denfivontinib) 150mg QD (Experimental): Administered orally
  Interventions: Drug: SKI-G-801
- SKI-G-801(Denfivontinib) 225mg QD (Experimental): Administered orally
  Interventions: Drug: SKI-G-801
- SKI-G-801(Denfivontinib) 300mg QD (Experimental): Administered orally
  Interventions: Drug: SKI-G-801
- SKI-G-801(Denfivontinib) 400mg QD (Experimental): Administered orally
  Interventions: Drug: SKI-G-801
- SKI-G-801(Denfivontinib) 500mg QD (Experimental): Administered orally
  Interventions: Drug: SKI-G-801

INTERVENTIONS:
Drug: SKI-G-801 — Oral SKI-G-801(Denfivontinib) will be daily administered based on dose level.
  Other Names: Denfivontinib

SUMMARY:
This is a phase I study intended to determine the MTD and RP2D of SKI-G-801 monotherapy by assessing the safety and tolerability including dose-limiting toxicity (DLT) at various dose levels and to explore the efficacy and PK in patients with advanced solid tumors.

DETAILED DESCRIPTION:
This is an open-label, monotherapy study in patients with advanced solid tumors, to evaluate the safety, tolerability, and pharmacokinetics (PK) of multiple ascending doses of SKI-O-801(Denfivontinib). A total of 36 subjects are planned to participate in 6 cohorts (traditional 3+3 design). In each cohort, 3 subjects will receive SKI-O-801. Dosing will be initiated with a 100 mg once daily (QD) dose cohort and escalated to 500 mg QD. After 1 cycle (28 days) of treatment if 3 subjects in each cohort have no DLT(Dose Limiting Toxicity), escalate the next dose level by Safety Review Committee decision.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults aged 19 years and older
* Subjects with histologically and/or cytologically confirmed, unresectable advanced or metastatic solid tumors that are confirmed as PD after the standard of care currently known to have clinical benefits, or for which no currently available standard therapies exist due to intolerance, ineligibility, refusal, etc.
* At least 1 evaluable lesion based on RECIST version 1.1 (the irradiated area or biopsied lesion will be considered evaluable if PD is demonstrated).
* The Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0-1
* Life expectancy of at least 12 weeks
* The last screening test results obtained within 7 days prior to the first dose of the IP (baseline) meet the following (with no administration of granulocyte colony-stimulating factor [G-CSF] or erythropoietin [EPO], or transfusion within 14 days prior to the laboratory tests)

  1. Hematological function ANC ≥1,500/μL Hemoglobin ≥9 g/dL Platelet count ≥100,000/μL
  2. Renal function: Creatinine clearance (CrCl) ≥45 mL/min (MDRD equation)
  3. Hepatic function AST ≤2.0 × ULN ALT ≤2.0 × ULN (AST/ALT ≤5 × ULN, if hepatic metastasis is confirmed) Total bilirubin ≤1.5 × ULN (<3.0 × ULN, if Gilbert's syndrome is confirmed)
  4. Blood coagulation function: prothrombin time (PT) (international normalized ratio [INR]) and activated partial thromboplastin time (aPTT) ≤1.5 × ULN (with an exception of PT or aPTT in the therapeutic range as per the purpose of anticoagulants if the subject is taking anticoagulants such as warfarin, heparin, or low molecular weight heparin)
* Voluntary written consent to participate in this study

Exclusion Criteria:

* 7th line or greater palliative systemic anti-cancer therapy for advanced or metastatic solid tumors (postoperative adjuvant therapy is considered as a single line of therapy if the disease recurs within 6 months after the last treatment, while endocrine therapy is excluded from the line of therapy)
* History of AXL inhibitors
* Difficulty (e.g., problem swallowing) in oral administration of SKI-G-801 or disease (celiac disease, Crohn's disease, or intestinal resection which is clinically significant or impacts absorption) which impact absorption
* Hypersensitivity to the active ingredient or excipients of SKI-G-801
* Major surgery within 4 weeks prior to IP administration
* Minor surgery within 2 weeks prior to IP administration
* Women who have a positive pregnancy test or are pregnant or breastfeeding at screening, or female subjects of childbearing potential or male subjects who do not agree to remain abstinent or use effective methods of contraception** for at least 27 weeks (female subjects) or 14 weeks (male subjects) after the last dose of the IP

  **Effective forms of contraception are defined as the following:
  1. Hormonal contraceptives (implants, injectables, oral contraceptives, etc.)
  2. Intrauterine device or intrauterine system (copper loop, hormone containing intrauterine system)
  3. Surgical sterilization (vasectomy, tubal ligation, etc.) of a subject or spouse (or partner)
  4. Double-barrier method with spermicide (including condom, diaphragm, vaginal sponge, or cervical cap; a male and a female condom must not be used together)
* Toxicity associated with prior anti-cancer therapy that does not resolve to Grade ≤1 or baseline (with the exceptions of alopecia [any grade], Grade ≤2 neuropathy, and endocrinopathy that is not controlled by hormone replacement therapy)
* History of using another investigational product/device within 4 weeks (or 5 half-lives, whichever is shorter) prior to IP administration
* Ineligibility or inability to participate in the study at the judgement of the investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-01-25 (Actual); Primary Completion 2024-04-23 (Estimated); Study Completion 2024-10-04 (Estimated)

PRIMARY OUTCOMES:
Determination of the MTD and/or RP2D based on DLTs | Study Day 1 up to Day 28 (each cycle is 28 days)
  For DLTs, the number of subjects, incidence, and number of events will be presented by dose group
The number of treatment discontinuation or dose reduction | Approximately 2 year
  The number of treatment discontinuation or dose reduction due to ADRs(Adverse Drug Reactions) will be presented by dose group.
AEs(Adverse event) | Approximately 2 year
  The number of AEs, the number of subjects affected, and the incidence will be presented.
Laboratory tests | Approximaely 8 weeks
  The number of participants with abnormal Laboratory test results such as hematology and chemistry lab results.

SECONDARY OUTCOMES:
Cmax | Approximately 29 days (Up to Cycle 2 Day 1)
  Maximum Plasma Concentration of SKI-G-801
AUC | Approximately 29 days (Up to Cycle 2 Day 1)
  Area under the plasma concentration versus time curve of SKI-G-801
Objective Response Rate (ORR) | Approximately 2 year
  The frequency and percentage of ORR will be presented by dose group using best overall response (BOR) based on RECIST version 1.1

CONTACTS AND LOCATIONS:
Locations (3):
- South Korea (3):
  - Yonsei University College of Medicine Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul